CLINICAL TRIAL: NCT04269473
Title: Evaluation of a Video Telehealth Gait Retraining Program Versus a Standard Exercise and Education Program for Patients With Running-Related Knee Pain
Brief Title: Video Telehealth Gait Retraining for Running-Related Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RHC-A-19-035; 19KACH004 (Other: Keller)
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Telemedicine; Running; Knee; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group will receive a telehealth gait retraining intervention in addition to standard physical therapy rehabilitation for running-related knee pain, which includes: an at-home exercise program, a return to running protocol, and standard physical therapy evaluations.
  Interventions: Procedure: Telehealth Gait Retraining; Procedure: Standard Physical Therapy Treatment; Procedure: Return to Running Protocol; Procedure: At Home Exercise Program
- Control Group (Active Comparator): Participants in the control group will receive standard physical therapy rehabilitation for running-related knee pain, which includes: an at-home exercise program, a return to running protocol, and standard physical therapy evaluations.
  Interventions: Procedure: Standard Physical Therapy Treatment; Procedure: Return to Running Protocol; Procedure: At Home Exercise Program

INTERVENTIONS:
Procedure: Telehealth Gait Retraining — Telehealth gait retraining is a novel approach to train participants to adopt a non-rearfoot foot strike pattern during running via telecommunications. During telehealth gait retraining, video of a participant's running form are sent to clinicians over a mobile device app and running form feedback is given. This process is repeated once a week for four weeks and then every other week until week 8.
  Arms: Experimental Group
Procedure: Standard Physical Therapy Treatment — Participants receiving standard Physical Therapy will visit the Physical Therapy Clinic every 2 to 3 weeks to be treated by a Physical Therapist.
Procedure: Return to Running Protocol — The Return to Running protocol is a six-phase running volume progression to re-introduce running slowly and safely after experiencing a running-related injury.
Procedure: At Home Exercise Program — The At Home Exercise Program consists of 4 lower leg and foot exercises that participants can perform on their own time.

SUMMARY:
In this randomized control trial, participants with running-related knee pain will be randomly assigned to either an intervention group or a control group. Participants in the intervention group will receive a telehealth gait retraining intervention, an at-home exercise program, a return to running protocol, and standard physical therapy. Participants in the control group will receive an at-home exercise program, a return to running protocol, and standard physical therapy. Data will be collected before intervention, at 10-weeks, and at 14-weeks to determine efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty Soldier or Cadet between the ages of 18 to 60 years old
* Knee pain that occurs during and/or after running that was not due to a recent acute trauma (such as an accident or a fall) and that is a pain intensity of at least a '3' and no greater than a '7' on a numeric pain rating scale with '0' meaning "no pain" and '10' meaning the "worst possible pain"
* Fluent in speaking and reading English

Exclusion Criteria:

* Currently on an Army running limiting profile for something other than knee pain
* Presence of rheumatoid or neurological diseases
* Plans to deploy or permanent change of station (PCS) within 4 months
* Current lower extremity injury other than knee pain
* History of traumatic knee injury (such as a surgery, ligament tear, or meniscal tear)
* Current pregnancy
* Inability to perform 20 unassisted single leg heel raises on each leg
* A non-rearfoot strike pattern during running
* Showing signs of ligamentous instability, meniscus pathology, or knee effusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Worst knee pain during running assessed by Visual Analogue Scale (VAS) | Change from baseline to 10-weeks
  Worst knee pain intensity in the past 7 days recorded using a 0 to 10 cm visual analogue scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Worst knee pain after running assessed by Visual Analogue Scale (VAS) | Change from baseline to 10-weeks
  Worst knee pain intensity in the past 7 days recorded using a 0 to 10 cm visual analogue scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Foot strike pattern during running measured with motion capture | Change from baseline to 10-weeks
  Portion of the foot that makes initial contact with the ground at the start of each stance phase during running.

SECONDARY OUTCOMES:
University of Wisconsin Running Injury and Recovery Index | Change from baseline to 10-weeks and 14-weeks
  A 9-item questionnaire (range 0-36, higher scores indicate more function) that measures a runners assessment of running ability after sustaining a running-related injury.
Worst non-knee pain during running assessed by Visual Analogue Scale (VAS) | Change from baseline to 10-weeks and 14-weeks
  Worst pain intensity in a region other than the knee during running in the past 7 days recorded using a 0 to 10 cm visual analogue scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Worst knee pain overall assessed by Visual Analogue Scale (VAS) | Change from baseline to 10-weeks and 14-weeks
  Worst knee pain intensity experienced overall in the past 7 days recorded using a 0 to 10 cm visual analogue scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Knee function assessed with the single assessment numeric evaluation method | Change from baseline to 10-weeks and 14-weeks
  Participants will rate their knee function on a scale of 0 (least normal) to 100 (most normal).
Knee function assessed with the anterior knee pain scale | Change from baseline to 10-weeks and 14-weeks
  Participants will rate their level of pain, disability, and impairment associated with their knee injury using a 13-item questionnaire (range 0-100, higher scores indicate better function).
Worst knee pain during running assessed by Visual Analogue Scale (VAS) | Change from baseline to 14-weeks
  Worst knee pain intensity in the past 7 days recorded using a 0 to 10 cm visual analogue scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Worst knee pain after running assessed by Visual Analogue Scale (VAS) | Change from baseline to 14-weeks
  Worst knee pain intensity in the past 7 days recorded using a 0 to 10 cm visual analogue scale where 0 equals no pain and 10 indicates the most severe pain the patient could imagine. Higher numbers equal greater levels of reported pain.
Foot strike pattern during running measured with motion capture | Change from baseline to 14-weeks
  Portion of the foot that makes initial contact with the ground at the start of each stance phase during running.

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital - Arvin Physical Therapy, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crowell MS, Brindle RA, Miller EM, Reilly N, Ford KR, Goss DL. The effectiveness of telehealth gait retraining in addition to standard physical therapy treatment for overuse knee injuries in soldiers: a protocol for a randomized clinical trial. Trials. 2023 Oct 16;24(1):672. doi: 10.1186/s13063-023-07502-x. PMID 37845752

DOCUMENTS (1):
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT04269473/ICF_000.pdf